CLINICAL TRIAL: NCT04728217
Title: Health Related Quality of Life of Youth and Young Adults With Haemophilia A Treated With Efmoroctocog Alfa in Russia
Brief Title: Health Related Quality of Life of Youth and Young Adults With Haemophilia A
Acronym: RELOQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The League of Clinical Research, Russia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RELOQ
Record Dates: First submitted 2021-01-20; First posted 2021-01-28 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Hemophilia A
Keywords: Haemophilia A; Health-related Quality of Life; Efmoroctocog alfa
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Intervention Model Description: A 12-month prospective open-label, single-arm multicentre study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients receiving Efmoroctocog alfa (Experimental): For long term prophylaxis, the recommended starting dose is 50 IU of factor VIII per kg body weight at intervals of 3 to 5 days. The dose may be adjusted based on patient response in the range of 25 to 65 IU/kg. In some cases, especially in younger patients, shorter dosage intervals or higher doses may be necessary.
  Interventions: Drug: Efmoroctocog Alfa Injection [Eloctate]

INTERVENTIONS:
Drug: Efmoroctocog Alfa Injection [Eloctate] — Efmoroctocog alfa should be administered according to Summary of Product Characteristics (SmPC)/ Instruction on Medical Use approved by Russian Ministry of Health ЛП-006034 (13.01.2020).

SUMMARY:
Research question:

Whether there are the changes in quality of life in patients with haemophilia A after switching from SHL FVIII prophylaxis to efmoroctocog alfa prophylaxis?

A 12-month prospective open-label, single-arm multicentre study. Evaluation of parameters will be carried out on the backdrop of patient treatment in the settings of routine medical practice. No medical examinations/ procedures/ treatment(s) on the top of regular medical practice are planned, except fixed time of examinations.

DETAILED DESCRIPTION:
Quality of life is among the key factors when medical decision about management of haemophilia is taken. There are no scientific data on the HRQoL in patients after switching from Standard Half Life (SHL) FVIII prophylaxis to efmoroctocog alfa (Extended Half Life, EHL) prophylaxis in Russia.

It will be a 12-month prospective open-label, single-arm multicentre study. Evaluation of parameters will be carried out on the backdrop of patient treatment in the settings of routine medical practice. No medical examinations/ procedures/ treatment(s) on the top of regular medical practice are planned, except fixed time of examinations. Providing the centers/ patients with the study drug (efmoroctocog alfa) may be considered as interventional component, whereas all administrations should be in accordance with Instruction on Medical Use approved by Russian Ministry of Health.

Research question:

Whether there are the changes in quality of life in patients with haemophilia A after switching from SHL FVIII prophylaxis to efmoroctocog alfa prophylaxis?

No hypothesis is formulated for this exploratory study. The obtained data will be used to assess real world data on quality of life and clinical outcomes in patients with haemophilia A after switching from SHL FVIII prophylaxis to efmoroctocog alfa prophylaxis in routine medical practice in Russia

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent form.
2. Adults, adolescents and children (12-25 years old) with haemophilia A with ABR ≥ 2 on at least one-year SHL FVIII prophylaxis.

Exclusion Criteria:

1. Patients who have had hypersensitivity reactions to efmoroctocog alfa or other constituents of the product.
2. History of Factor VIII inhibitors.
3. Patients who have other haemostatic disorders.
4. Patients participating in interventional studies.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Health-related quality of life | Month 12
  Haemophilia Adult Quality of Life Questionnaire (Haem-A-QoL) - for patients of 18-25 y.o.; total score, domain scores.
  or Haemophilia-specific Quality of Life assessment for children and adolescents Short Form (Haemo-QoL SF) - for patients 12-17 y.o.; total score, domain scores.

SECONDARY OUTCOMES:
Spontaneous bleedings | Month 1 - Month 3 - Month 6 - Month 12
  Number from previous visit
Spontaneous bleedings - localisation | Month 1 - Month 3 - Month 6 - Month 12
  Localisation of spontaneous bleedings: joints, muscles, subcutaneous/ submucosal, abdominal/ gastrointestinal, retroperitoneal, genitourinary, CNS, pharyngeal, other.
Post-traumatic bleedings | Month 1 - Month 3 - Month 6 - Month 12
  Number from previous visit
Post-traumatic bleedings - localisation | Month 1 - Month 3 - Month 6 - Month 12
  Localisation of post-traumatic bleedings: joints, muscles, subcutaneous/ submucosal, abdominal/ gastrointestinal, retroperitoneal, genitourinary, CNS, pharyngeal, other.
Administration of efmorococtog alfa for correction of bleedings | Month 1 - Month 3 - Month 6 - Month 12
  Dose of efmorococtog alfa: IU.
Surgery/ Invasive Procedures: major | Month 1 - Month 3 - Month 6 - Month 12
  Number from previous visit.
Surgery/ Invasive Procedures: minor | Month 1 - Month 3 - Month 6 - Month 12
  Number from previous visit.
Administration of efmorococtog alfa for correction of bleedings for Surgery/ Invasive Procedures | Month 1 - Month 3 - Month 6 - Month 12
  Dose of efmorococtog alfa: IU.
Hospitalisations | Month 1 - Month 3 - Month 6 - Month 12
  Number from previous visit.
Hospitalisations: duration | Month 1 - Month 3 - Month 6 - Month 12
  Total duration of all hospitalisations: days.
Hemophilia Joint Health Score | Day 0 - Month 6 - Month 12
  Hemophilia Joint Health Score 2.1 for knee, elbow, ankle (left, right): score.
Target Joints | Day 0 - Month 6 - Month 12
  Target joints: knee, elbow, ankle, hip, shoulder, carpal, other (left, right): yes/ no.
Ultrasound Scoring | Day 0 - Month 6 - Month 12
  Ultrasound scoring (HEAD-US): score.
Factor VIII Activity | Day 0 - Month 1 - Month 3 - Month 6 - Month 12
  Factor VIII Activity (before injection; 30 min after injection), clotting assays (one stage): IU/dL.
Factor VIII Inhibitor Activity | Day 0 - Month 1 - Month 3 - Month 6 - Month 12
  Factor VIII Inhibitor Activity: Nijmegen-Bethesda unit/mL.
Administration of efmoroctocog alfa | Day 0 - Month 1 - Month 3 - Month 6 - Month 12
  Administration of efmoroctocog alfa, frequency: no. of injections per week.
Administration of efmoroctocog alfa: factor consumption | Day 0 - Month 1 - Month 3 - Month 6 - Month 12
  Administration of efmoroctocog alfa, factor consumption: IU per week, IU/kg per week (calculation).
Previous treatment/ prophylaxis of haemophilia | Day 0 - Month 1 - Month 3 - Month 6 - Month 12
  Generic drug name.

CONTACTS AND LOCATIONS:
Locations (1):
- League of Clinical Research (LeagueCRR), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No